CLINICAL TRIAL: NCT05450510
Title: Effects of Slow and Accelerated Rehabilitation Protocols After Latissimus Dorsi Transfer in Massive, Irreparable Rotator Cuff Tears
Brief Title: Slow and Accelerated Rehabilitation Protocols
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022500
Record Dates: First submitted 2022-06-30; First posted 2022-07-08 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Injuries; Rotator Cuff Tears; Pain, Shoulder
Keywords: Rotator Cuff Injuries; tear; pain; shoulder
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Lacerations; Pain | interventions — Acceleration

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Masking Description: blinded assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Accelerated (ACCEL) physiotherapy group (Active Comparator): They will be referred to Physiotherapy and Rehabilitation clinics for a 8-week-long Phase 2 and Phase 3 trainings. The training program includes the following exercises: cold-pack ; TENS (60-120 Hz); soft tissue massage, joint mobilizations; mobility exercises; stretching, controlled strengthening and endurance exercises.
  Interventions: Other: Accelerated (ACCEL) protocol group
- Slow (SLOW) physiotherapy group (Active Comparator): They will be referred to Physiotherapy and Rehabilitation clinics for a 14-week-long Phase 2 and Phase 3 trainings. The training program includes the following exercises: cold-pack ; TENS (60-120 Hz); soft tissue massage, joint mobilizations; mobility exercises; stretching, controlled strengthening and endurance exercises.
  Interventions: Other: Slow (SLOW) protocol group

INTERVENTIONS:
Other: Accelerated (ACCEL) protocol group — After randomization and initial evaluations, patients will be referred to Physiotherapy and Rehabilitation clinics for a 8-week-long Phase 2 and Phase 3 trainings.
  Arms: Accelerated (ACCEL) physiotherapy group
Other: Slow (SLOW) protocol group — After randomization and initial evaluations, patients will be referred to Physiotherapy and Rehabilitation clinics for a 14-week-long Phase 2 and Phase 3 trainings.
  Arms: Slow (SLOW) physiotherapy group

SUMMARY:
Latissimus dorsi transfer is an established treatment option with favorable results in massive, irreparable rotator cuff tears, however, it is controversial if earlier motion is detrimental or beneficial to the postoperative goal of reduced pain and improved clinical outcomes. Therefore, the aim of this study is to compare the effects of slow and accelerated rehabilitation protocols after latissimus dorsi transfer in massive, irreparable rotator cuff tears.

DETAILED DESCRIPTION:
A variety of surgical options are proposed in the treatment of massive cuff tears. The treatment options include acromioplasty and tuberoplasty, partial repair with or without soft tissue augmentation, latissimus dorsi transfer (LDT), superior capsular reconstruction (SCR), and reverse total shoulder arthroplasty. Among these options, LDT is a well-recognized technique that aims to rebalance the soft tissue tension around the shoulder joint in order to prevent superior escape of the humeral head and loss of function. From a biomechanical standpoint, the transferred tendon is theorized to function as a humeral head depressor by means of a tenodesis effect, as well as by increasing the active external rotation through the transfer vector. It is an established treatment option with favorable results, however, it is controversial if earlier motion is detrimental or beneficial to the postoperative goal of reduced pain and improved clinical outcomes. Therefore, the aim of this study is to compare the effects of slow and accelerated rehabilitation protocols after latissimus dorsi transfer in massive, irreparable rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

* being in the age range of 18-65 years
* being diagnosed with massive, irreparable rotator cuff tears based on magnetic resonance imaging and clinical continuity tests
* symptoms are unresponsive to conservative care including steroid injections and physiotherapy for at least 6 months
* having a good command of the Turkish language
* scoring above 24 in the Mini Mental State Test
* ≥80% compliance in completing the post-ARCR Phase 1 trainings
* volunteering to participate in the study

Exclusion Criteria:

* diabetes mellitus
* neurological problems
* cervical disc herniation
* visual, verbal, and/or cognitive defects (aphasia, unilateral neglect, etc.)
* systemic inflammatory problems
* hypermobility, trauma, and/or inflammation that could be a contraindication for mobilization
* former shoulder fractures on the affected side
* advanced glenohumeral arthritis (Hamada grade 3),
* deltoid muscle dysfunction,
* irreparable subscapularis tears,
* active infection,
* shoulder stiffness,
* a history of previous shoulder surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 14 weeks
  Visual analog scale is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
The Disabilities of the Arm, Shoulder and Hand Questionnaire | 14 weeks
  The Disabilities of the Arm, Shoulder and Hand Questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. It consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
American Shoulder and Elbow Surgeons score | 14 weeks
  It is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points. Patients can complete the questionnaire in less than five minutes. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Western Ontario Rotator Cuff Index | 14 weeks
  It has 21 items in four domains, including physical symptoms (ten questions), sports/recreation/work (four questions), lifestyle (four questions) and emotions (three questions). Raw scores range from 0 to 2100 with a higher score indicating decreased quality of life due to pathological condition of the rotator cuff. Mathematic conversion yields a percentage score; higher percentages indicate proximity to normal function.
Constant-Murley Shoulder Score | 14 weeks
  Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively. In the original publication, the pain experienced during normal activities of daily living was scored as: no pain = 15 points, mild = 10, moderate = 5 and severe = 0 points.

SECONDARY OUTCOMES:
Catastrophizing | 14 weeks
  Pain Catastrophizing Scale will be used to evaluate the patient's feelings, thoughts, and emotions related to cognitive characteristics of pain. It is a self-administered questionnaire with 13 items and 3 subscales: helplessness, magnification, and rumination. A 5-point scale is used for each item, with higher values representing greater catastrophizing. The scores for each item are added to determine the subscales, and the total score is calculated by the summation of all items. The PCS scores range from 0 to 52 points.
Hospital Anxiety and Depression Scale | 14 weeks
  It will be used to assess anxiety and depression. It consists of 7 items for anxiety and 7 for depression. The items are scored on a 4-point scale from 0 (not present) to 3 (considerable).
Tampa-Scale of Kinesiophobia | 14 weeks
  Participants will be assessed with Tampa-Scale of Kinesiophobia in terms of presence of kinesiophobia. The TSK is a 17-item scale that measures the somatic focus of patients (beliefs about underlying and serious medical problems), and activity avoidance (beliefs about (re) injury or increased pain). The TSK has moderate construct, concurrent and predictive validity, good internal consistency, and a moderate to good retest reliability. Patients scoring high on the TSK, above 37 points, are likely to have fear of movement.
12-Item Short-Form Health Survey | 14 weeks
  Participants will be assessed with 12-Item Short-Form Health Survey in terms of quality of life. It is a self-administered survey and two scores can be measured: the Physical Component and the Mental Component. In both, scores range from 0 to 100, with the highest scores associated with better levels of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozturk BY, Ak S, Gultekin O, Baykus A, Kulduk A. Prospective, randomized evaluation of latissimus dorsi transfer and superior capsular reconstruction in massive, irreparable rotator cuff tears. J Shoulder Elbow Surg. 2021 Jul;30(7):1561-1571. doi: 10.1016/j.jse.2021.01.036. Epub 2021 Mar 4. PMID 33675971
- [Background] Anastasopoulos PP, Alexiadis G, Spyridonos S, Fandridis E. Latissimus Dorsi Transfer in Posterior Irreparable Rotator Cuff Tears. Open Orthop J. 2017 Feb 28;11:77-94. doi: 10.2174/1874325001711010077. eCollection 2017. PMID 28400877
- [Background] Burnier M, Lafosse T. Pectoralis Major and Anterior Latissimus Dorsi Transfer for Subscapularis Tears. Curr Rev Musculoskelet Med. 2020 Dec;13(6):725-733. doi: 10.1007/s12178-020-09674-4. PMID 32833188
- [Background] Elhassan BT, Wagner ER, Kany J. Latissimus dorsi transfer for irreparable subscapularis tear. J Shoulder Elbow Surg. 2020 Oct;29(10):2128-2134. doi: 10.1016/j.jse.2020.02.019. Epub 2020 Jun 9. PMID 32573448
- [Background] Wieser K, Ernstbrunner L, Zumstein MA. Surgical Management of Massive Irreparable Cuff Tears: Latissimus Dorsi Transfer for Posterosuperior Tears. Curr Rev Musculoskelet Med. 2020 Oct;13(5):605-611. doi: 10.1007/s12178-020-09659-3. PMID 32661917
- [Background] Galasso O, Mantovani M, Muraccini M, Berardi A, De Benedetto M, Orlando N, Gasparini G, Castricini R. The latissimus dorsi tendon functions as an external rotator after arthroscopic-assisted transfer for massive irreparable posterosuperior rotator cuff tears. Knee Surg Sports Traumatol Arthrosc. 2020 Jul;28(7):2367-2376. doi: 10.1007/s00167-019-05819-2. Epub 2019 Dec 6. PMID 31811355